CLINICAL TRIAL: NCT07321769
Title: Full 3D Eye Modeling in the Diagnosis and Treatment of Lens Diseases With Eye Structures Disorders
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1229
Record Dates: First submitted 2025-12-07; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Lens Diseases
MeSH Terms: conditions — Lens Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Toward 3D Modeling for Lens Disorders Associated with Congenital Anomalies: Part I: Exploration and research on full three-dimensional modeling in the diagnosis and treatment of lens diseases with congenital developmental anomaliesa
- Toward 3D Modeling for Reconstructive Management of Ocular Trauma: Part II: Exploration and research on full three-dimensional modeling for the reconstruction and treatment of ocular trauma
- Toward 3D Modeling for IOL Spatial Positioning: Part III: Exploration and research on full three-dimensional modeling for the spatial positioning of pseudophakic eyes
- Toward 3D Modeling for Cataracts with Iris/Pupillary Abnormalities: Part IV: Exploration and research on full three-dimensional modeling for cataract patients with iris or pupillary abnormalities
- Toward 3D Modeling for Cataracts with Posterior Segment Diseases: Part V: Exploration and research on full three-dimensional modeling for the management and treatment of cataract patients with posterior segment diseases
- Normal Control Group: Exploration and research on full three-dimensional modeling for individuals with no significant structural ocular diseases served as the normal control group.

SUMMARY:
In patients with complex cataracts, spatial abnormalities in the lens and its surrounding tissues-including both the anterior and posterior ocular segments-are often present. Due to the lack of precise preoperative assessment tools and standardized surgical protocols, these cases are associated with increased surgical complexity and difficulty, often leading to suboptimal visual outcomes. Therefore, this study explores a three-dimensional reconstruction method for the anterior segment based on swept-source optical coherence tomography (SS-OCT). By integrating imaging data from CT, B-scan ultrasound, and ultrasound biomicroscopy (UBM), a full three-dimensional model of the eye is constructed to enable objective and quantitative evaluation of its entire structure. This approach aims to provide valuable reference for surgical planning and prognostic assessment in lens diseases accompanied by ocular spatial structural abnormalities.

DETAILED DESCRIPTION:
In patients with complex cataracts, lens opacities are often accompanied by spatial structural disorders or abnormalities involving both the lens itself and its surrounding tissues, including the anterior and posterior ocular segments. Due to the lack of precise preoperative assessment tools and standardized surgical protocols, these cases present higher surgical complexity and technical difficulty, often resulting in suboptimal outcomes. Therefore, preoperative objective quantitative analysis of the three-dimensional morphology and spatial relationships of the anterior segment, posterior segment, and the entire globe is crucial for surgical planning, prevention of complications, and postoperative visual recovery.

This study employs a retrospective research design. Using multimodal imaging systems-including anterior segment swept-source optical coherence tomography (SS-OCT), CT, B-scan ultrasound, and ultrasound biomicroscopy (UBM)-we aim to explore methods for full-eye three-dimensional reconstruction. The goal is to construct a comprehensive 3D ocular model that includes the cornea, anterior chamber, iris, angle, lens, vitreous cavity, retina, and related fundus structures.

This model will be used to comprehensively analyze morphological and spatial alterations in lens diseases associated with ocular spatial abnormalities, providing an objective quantitative description. Furthermore, the study will validate the effectiveness of this full 3D ocular model in clinical diagnosis, surgical planning, and prognosis assessment for this broad category of conditions. Ultimately, it seeks to establish objective, quantitative reference standards for the precise diagnosis and treatment of lens diseases complicated by ocular spatial structural disorders.

ELIGIBILITY:
Inclusion Criteria:

* Part I：Toward 3D Modeling for Lens Disorders Associated with Congenital Anomalies

  1) Diagnosed with lens disorders such as lens subluxation or deformity via imaging (slit-lamp, UBM) or clinical examination, combined with conditions such as megalocornea, microcornea, nanophthalmos, keratoconus, or iris coloboma; 2) Presence of imageable ocular structures; 3) Able to cooperate with and complete relevant examinations including B-scan ultrasound, UBM, and anterior segment SS-OCT.
* Part II: Toward 3D Modeling for Reconstructive Management of Ocular Trauma 1) Diagnosed with previous or stabilized corneal trauma, traumatic cataract, or iris injury, with or without associated vitreous traction or retinal damage; 2) Patients with open globe injuries that have been managed, with closed wounds and no endophthalmitis; 3) Able to cooperate with and complete relevant examinations including B-scan ultrasound, UBM, anterior segment SS-OCT, and CT.
* Part III:Toward 3D Modeling for IOL Spatial Positioning 1) Patients who have undergone cataract extraction with intraocular lens (IOL) implantation (in-the-bag or scleral-fixated); 2) Stable IOL position post-implantation with clear documentation of IOL parameters; 3) Able to cooperate with and complete relevant examinations including B-scan ultrasound, UBM, and anterior segment SS-OCT.
* Part IV: Toward 3D Modeling for Cataracts with Iris/Pupillary Abnormalities

  1. Patients with iris morphological or positional abnormalities due to previous uveitis, trauma, or developmental anomalies (e.g., iris atrophy, synechiae, iridodialysis, polycoria, pupillary membrane remnants); 2) Able to cooperate with and complete relevant examinations including B-scan ultrasound, UBM, and anterior segment SS-OCT.
* Part V: Toward 3D Modeling for Cataracts with Posterior Segment Diseases

  1) Patients with various posterior segment vitreoretinal diseases (e.g., vitreous traction or proliferation, macular hole, epiretinal membrane), with or without anterior segment spatial structural abnormalities; 2) Able to cooperate with and complete relevant examinations including B-scan ultrasound, UBM, and anterior/posterior segment SS-OCT.
* Part VI: Normal Control Group

  1. No significant structural ocular diseases; 2) Healthy fellow eyes of unilateral ocular trauma patients from Part II, with no notable anterior or posterior segment abnormalities; 3) Able to cooperate with and complete relevant examinations including B-scan ultrasound, UBM, anterior/posterior segment SS-OCT, and CT.

Exclusion Criteria:

* Part I: Toward 3D Modeling for Lens Disorders Associated with Congenital Anomalies

  1) Concurrent open globe injury or severe ocular deformity; 2) Excessive corneal opacity or severe edema resulting in inadequate image quality; 3) Severe dry eye or tear film abnormalities affecting imaging;4) Severe ocular structural deformity preventing effective 3D model reconstruction; 5) Severe systemic disease precluding tolerance of the examination; 6) Contraindications to B-scan ultrasound or UBM, conditions impairing imaging, or allergy to coupling gel.
* Part II: Toward 3D Modeling for Reconstructive Management of Ocular Trauma

  1) Unmanaged open globe injury or severe ocular deformity; 2) Severe systemic disease precluding tolerance of the examination; 3) Contraindications to CT imaging (e.g., metallic implants in the head/face region, pregnancy, lactation) or history of contrast medium allergy/adverse reactions.
* Part III: Toward 3D Modeling for IOL Spatial Positioning

  1) Unclear IOL position or documented implantation failure; 2) Corneal opacity or severe pupillary abnormality affecting imaging; 3) IOL instability due to intra- or postoperative complications preventing imaging;4) Open globe injury or severe ocular deformity; 5) Severe systemic disease precluding tolerance of the examination; 6) Contraindications to B-scan ultrasound or UBM, conditions impairing imaging, or allergy to coupling gel.
* Part IV: Toward 3D Modeling for Cataracts with Iris/Pupillary Abnormalities

  1) Corneal opacity or hyphema preventing imaging; 2) Severe global ocular deformity precluding imaging; 3) Severe systemic disease precluding tolerance of examination or follow-up; 4) Contraindications to B-scan ultrasound or UBM, conditions impairing imaging, or allergy to coupling gel.
* Part V: Toward 3D Modeling for Cataracts with Posterior Segment Diseases

  1) Severe structural deformity of both anterior and posterior segments preventing effective 3D model reconstruction; 2) Severe systemic disease precluding tolerance of examination or follow-up; 3) Contraindications to B-scan ultrasound or UBM, conditions impairing imaging, or allergy to coupling gel.
* Part VI: Normal Control Group 1) History of severe ocular trauma or ocular surgery; 2) Conditions affecting imaging quality, including corneal opacity, severe dry eye, tear film abnormalities, anterior segment disease, or significant retinal pathology; 3) Severe systemic disease precluding tolerance of the examination; 4) Contraindications to CT imaging (e.g., metallic implants in the head/face region, pregnancy, lactation) or history of contrast medium allergy/adverse reactions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The data for this project was collected from patients who visited the Second Affiliated Hospital, School of Medicine, Zhejiang University from January 1, 2020 to December 31, 2025.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anterior Segment SS-OCT Quantitative Results | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Quantification of the anterior segment SS-OCT imaging results
Computed tomography | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Quantification of ocular CT imaging results
B-scan ultrasonography | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Quantification of the B-ultrasound imaging results of the eyes
Ultrasound Biomicroscope | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Quantification of the results of ocular UBM examination

SECONDARY OUTCOMES:
IOL tilt decentration ELP | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Using SS-OCT to record the effective position of the IOL.
Surgical Record | During the operation
  Intraoperative documentation included surgical procedures, irrigation system parameters, phacoemulsification energy, and other relevant information.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Phd, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine,, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided